CLINICAL TRIAL: NCT02814123
Title: A Randomized, Three-way, Crossover Study to Assess the Efficacy of Fast-acting Insulin-plus-pramlintide Closed-loop Co-administration, Regular Insulin-plus-pramlintide Closed-loop Co-administration, and Fast-acting Insulin-alone Closed-loop Infusion in Regulating Glucose Levels Over a 24-hour Period in Adults With Type 1 Diabetes in Inpatient Settings.
Brief Title: Effect of Basal-Bolus Closed-Loop Co-Administration of Insulin and Pramlintide on Improving the Glycemic Control in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Ahmad Haidar, Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAP-1
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Pramlintide; Artificial Pancreas; Closed-Loop System; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rapid Insulin-alone closed-loop delivery (Active Comparator): Rapid Insulin will be delivered by subcutaneous infusion. Interventions: 24-hour inpatient intervention Drug: Rapid acting Insulin (aspart, lispro, glulisine)
  Interventions: Other: 24-hour inpatient intervention
- Rapid Insulin-plus-pramlintide closed-loop delivery (Experimental): Rapid insulin and pramlintide will be delivered by subcutaneous infusion using a fixed ratio (6 µg pramlintide/unit insulin).
  Interventions: 24-hour inpatient intervention Drug: Rapid acting Insulin (aspart, lispro, glulisine) Drug: Pramlintide
  Interventions: Other: 24-hour inpatient intervention
- Regular Insulin-plus-pramlintide closed-loop delivery (Experimental): Regular insulin and pramlintide will be delivered by subcutaneous infusion using a fixed ratio (6 µg pramlintide/unit insulin).
  Interventions: 24-hour inpatient intervention Drug: Regular Insulin (humulin R) Drug: Pramlintide
  Interventions: Other: 24-hour inpatient intervention

INTERVENTIONS:
Other: 24-hour inpatient intervention — Subjects will be admitted at the research facility at 7:30. A cannula will be inserted into an arm or a hand vein for blood sampling purposes. Each 24-hour intervention visit includes 3 standardized meals (8:00, 12:00, and 17:00), an evening snack (21:00) and an overnight stay. The glucose level as measured by the real time sensor will be entered manually into the computer every 10 minutes. The insulin and pramlintide pumps' infusion rates will then be changed manually based on the computer generated recommendation, while still maintaining the ratio. The computer generated recommendations are based on a predictive algorithm.

SUMMARY:
The closed-loop delivery system is composed of an insulin pump, a continuous glucose sensor and a dosing algorithm that calculates the insulin dose to infuse based on sensor readings. Pramlintide is a drug and an analog of amylin, a hormone that is co-secreted with insulin in healthy individuals, and is deficient in people with type 1 diabetes. Co-injection of pramlintide with insulin at meal times improves glucose control in type 1 diabetes. Literature data suggests that regular insulin may better match the effect of pramlintide compared to rapid insulin in regulating post-prandial glucose levels.

The purpose of this study is to compare the effectiveness of 3 strategies to control your day-and-night glucose levels:

1. rapid insulin-alone closed-loop delivery;
2. rapid insulin-plus-pramlintide closed-loop delivery;
3. regular insulin-plus-pramlintide closed-loop delivery.

The primary hypotheses are:

1. During closed-loop control, the simultaneous basal-bolus infusion of pramlintide and fast-acting insulin improves glucose control compared to fast-acting insulin-alone infusion.
2. During closed-loop control, the simultaneous basal-bolus infusion of pramlintide and regular insulin improves glucose control compared to fast-acting insulin-alone infusion.

DETAILED DESCRIPTION:
The closed-loop delivery system is composed of an insulin pump, a continuous glucose sensor and a dosing algorithm that calculates the insulin dose to infuse based on sensor readings. Pramlintide is a drug and an analog of amylin, a hormone that is co-secreted with insulin in healthy individuals, and is deficient in people with type 1 diabetes. Co-injection of pramlintide with insulin at meal times improves glucose control in type 1 diabetes.

Literature data suggests that the pharmacodynamics of regular insulin may better match the effect of pramlintide compared to the pharmacodynamics of fast-acting insulin. Moreover, the cost of regular insulin is significantly lower than fast-acting insulin. Therefore, if a similar (or better) glucose profile can be achieved with regular insulin-plus-pramlintide compared to fast-acting insulin-plus-pramlintide, then a co-formulation employing regular insulin should be prioritized.

Therefore, in this protocol, we aim to assess the effect of the simultaneous, closed-loop, basal-bolus infusion of pramlintide with insulin at a fixed ratio in controlling glucose levels. In the first experimental arm, we propose to infuse pramlintide with fast-acting insulin. In the second experimental arm, pramlintide will be infused with regular insulin. The control arm will be fast-acting insulin-alone closed-loop system.

The aim of the study is to assess the efficacy of the simultaneous, closed-loop, basal-bolus infusion of pramlintide with fast-acting insulin at a fixed ratio and pramlintide with regular insulin at a fixed ratio in controlling glucose levels compared to fast-acting insulin-alone closed-loop infusion.

The investigators aim to conduct a randomized, three-way, crossover trial to compare the efficacy of 1) fast-acting insulin-plus-pramlintide closed-loop delivery, 2) regular insulin-plus-pramlintide closed-loop delivery, and 3) fast-acting insulin-alone closed-loop delivery in regulating glucose levels over a period of 24 hours in a study on adults in inpatient settings. Insulin (fast-acting and regular) and pramlintide are given with fixed ratio (6 µg of pramlintide for each unit of insulin).

Before each 24-hour intervention visit, the participant's insulin therapy (basal rates and insulin-to-carbohydrate ratios) will be optimized for a minimum of 10 days, with a target of 14 days.

There will be a wash-out period of 0 to 42 days between the three intervention arms (termination of 24-hr intervention and start of next optimization period).

The primary hypotheses are:

1. During closed-loop control, the simultaneous basal-bolus infusion of pramlintide and fast-acting insulin improves glucose control compared to fast-acting insulin-alone infusion.
2. During closed-loop control, the simultaneous basal-bolus infusion of pramlintide and regular insulin improves glucose control compared to fast-acting insulin-alone infusion.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age.
* Clinical diagnosis of type 1 diabetes for at least 12 months. (The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.)
* The subject will have been on insulin pump therapy for at least 6 months.
* HbA1c ≤ 10%.

Exclusion Criteria:

* Current or ≤ 1 month use of other antihyperglycemic agents (SGLT2, GLP-1, Metformin, Acarbose, etc.…).
* Severe hypoglycemic episode within one month of screening.
* Severe diabetes keto-acidosis episode within one month of screening.
* Planned or ongoing pregnancy.
* Known or suspected allergy to the study drugs.
* Gastroparesis.
* Use of prokinetic drugs that stimulate gastric emptying (domperidone, cisapride, metoclopramide).
* Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
* Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
* Current use of glucocorticoid medication.
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
* Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
Percentage of time of plasma glucose levels spent in target range. Target range is defined to be between 3.9 and 10.0 mmol/L of fast-acting insulin-plus-pramlintide closed-loop delivery vs. fast-acting insulin-alone closed-loop delivery. | Up to 24 hours
Percentage of time of plasma glucose levels spent in target range. Target range is defined to be between 3.9 and 10.0 mmol/L of regular insulin-plus-pramlintide closed-loop delivery vs. fast-acting insulin-alone closed-loop delivery. | Up to 24 hours

SECONDARY OUTCOMES:
Percentage of time of plasma glucose levels spent in target range, comparing fast-acting insulin-plus-pramlintide closed-loop delivery vs. regular insulin-plus-pramlintide closed-loop delivery. | Up to 24 hours
Percentage of time (8:00-8:00) of plasma glucose levels spent: a. 3.9-7.8 mmol/L; b. 3.9-10 mmol/L; c. <3.9 mmol/L; d. <3.3 mmol/L; e. <2.8 mmol/L; f. >7.8 mmol/L; g. >10 mmol/L; h. >13.9 mmol/L; i. >16.7 mmol/L | Up to 24 hours
Percentage of overnight time (23:00-8:00) of plasma glucose levels: a. 3.9-7.8 mmol/L; b. 3.9-10 mmol/L; c. <3.9 mmol/L; d. <3.3 mmol/L; e. <2.8 mmol/L; f. >7.8 mmol/L; g. >10 mmol/L; h. >13.9 mmol/L; i. >16.7 mmol/L | Up to 24 hours
Standard deviation of glucose levels as a measure of glucose variability. | Up to 24 hours
Total insulin delivery. | Up to 24 hours
Total pramlintide delivery. | Up to 24 hours
Mean plasma glucose level during: a. the overall study period; b. overnight period. | Up to 24 hours
Mean plasma insulin concentration. | Up to 24 hours
Mean plasma glucagon concentration. | Up to 24 hours
Mean plasma amylin concentration. | Up to 24 hours
Number of subjects experiencing hypoglycemia requiring oral treatment during: a. the overall study period; b. the night. | Up to 24 hours
Gastrointestinal symptoms during the treatment optimization (i.e., the minimum 10 days prior to the 24-hour closed-loop visits) and during the 24-hour closed-loop visits. | Up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Haidar, Principal Investigator — McGill University; Laurent Legault, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haidar A, Tsoukas MA, Bernier-Twardy S, Yale JF, Rutkowski J, Bossy A, Pytka E, El Fathi A, Strauss N, Legault L. A Novel Dual-Hormone Insulin-and-Pramlintide Artificial Pancreas for Type 1 Diabetes: A Randomized Controlled Crossover Trial. Diabetes Care. 2020 Mar;43(3):597-606. doi: 10.2337/dc19-1922. Epub 2020 Jan 23. PMID 31974099
- [Derived] Tsoukas M, Rutkowski J, El-Fathi A, Yale JF, Bernier-Twardy S, Bossy A, Pytka E, Legault L, Haidar A. Accuracy of FreeStyle Libre in Adults with Type 1 Diabetes: The Effect of Sensor Age. Diabetes Technol Ther. 2020 Mar;22(3):203-207. doi: 10.1089/dia.2019.0262. Epub 2020 Jan 23. PMID 31613140

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02814123/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02814123/ICF_001.pdf